CLINICAL TRIAL: NCT01558414
Title: Prospective Randomized Clinical Trial Comparing Single Incision Laparoscopic Surgery vs Flexible Single Incision Surgery on Cholecystectomy
Brief Title: Single Incision Laparoscopic Surgery vs Flexible Single Incision Surgery for Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jose F. Noguera (Other)
Collaborators: Hospital Mateo Orfila (Other)
Responsible Party: Sponsor-Investigator, Jose F. Noguera, Chief Department of Surgery, Hospital Son Llatzer
Organization: Hospital Son Llatzer (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Llatzer-FSIS
Record Dates: First submitted 2012-03-17; First posted 2012-03-20 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Cholelithiasis; Surgery; Laparoscopy
Keywords: Cholecystectomy; Minimally invasive surgery; Laparoscopic surgery; Single incision surgery
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SILS (Experimental): Cholecystectomy performed by Single Incision Laparoscopic Surgery with the SILS TM device
  Interventions: Procedure: SILS Cholecystectomy
- FSIS (Experimental): Cholecystectomy performed by Flexible Single Incision Surgery with the flexible endoscope through a single incision at the umbilicus
  Interventions: Procedure: FSIS cholecystectomy
- Conventional laparoscopy (Active Comparator): Cholecystectomy performed by a conventional laparoscopic approach
  Interventions: Procedure: Conventional laparoscopy

INTERVENTIONS:
Procedure: SILS Cholecystectomy — Cholecystectomy performed by Single Incision Laparoscopic Surgery with the SILS TM device
  Arms: SILS
Procedure: FSIS cholecystectomy — Cholecystectomy performed by Flexible Single Incision Surgery with the flexible endoscope through a single incision at the umbilicus
  Arms: FSIS
Procedure: Conventional laparoscopy — Minimally invasive cholecystectomy through the conventional laparoscopic approach using 3 ports (one 11-cm umbilical port and two accessory 5-mm ports).
  Arms: Conventional laparoscopy

SUMMARY:
Prospective randomized pilot clinical trial, with 3 arms and one year follow up. The study will include 60 patients, with a 1:1:1 ratio, 20 patients per group. In 40 patients a transumbilical single site incision will be performed with two different manners: single-port device SILS TM (Single Incision Laparoscopic Surgery), and flexible endoscope and accessory trocars in a single incision (FSIS-Flexible Single Incision Surgery). The third group is the control one, a conventional laparoscopic approach.

The trial is designed as a pilot study to assess, as main objective, if these two endoscopic approaches have the same security and effectiveness in cholecystectomy.

Hypothesis:

Transumbilical approaches with single port and single incision with the flexible endoscope have the same efficacy and safety performing the endoscopic cholecystectomy.

Objectives:

Main objective:

Assess whether both approaches are equally safe in its application to endoscopic cholecystectomy.

Secondary objectives:

Investigate the differences in the rate of conversion to open surgery between different surgical approaches.

Investigate the differences in the rate of wound infection between the different surgical approaches.

Investigate the differences in the rate of postoperative incisional hernias between different surgical approaches.

Investigate whether there are differences in the rate of overall complications, all-cause mortality and the cost between different surgical approaches.

DETAILED DESCRIPTION:
Inclusion criteria:

* Patients affected with symptomatic cholelithiasis with elective surgical indication, not urgent, aged between 18 and 65.
* Signing of informed consent for cholecystectomy and specific consent for the trial.
* Anesthetic risk ASA I-II.

Exclusion criteria:

* Presence of acute cholecystitis and / or suspicion of occupation of the main bile duct.
* ASA III and higher.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 and under 65
* symptomatic cholelithiasis with an indication for laparoscopic surgery
* signed specific informed consent including specific information of the new surgical approach
* ASA 1 and 2.

Exclusion Criteria:

* current or previous cholecystitis
* current or previous suspected bile duct's problems
* previous abdominal surgery
* umbilical and other abdominal hernias
* some other condition with increased risk to infection or abdominal wall problems.
* ASA 3 and more

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Surgical safety | During surgical intervention
  Number of patients without clinical problems in the surgery

SECONDARY OUTCOMES:
Conversion to other surgical approach | During the surgical intervention
  Rate of conversion to conventional laparoscopic surgery and open surgery.

CONTACTS AND LOCATIONS:
Overall Officials: José F Noguera, MD, PhD, Study Director — Hospital Son Llàtzer; Juan C García, MD, Study Chair — Hospital Son Llàtzer
Locations (1):
- Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands, Spain

REFERENCES:
- [Background] Sanchez-Margallo FM, Perez FJ, Sanchez MA, Asencio JM, del Carmen Tejonero M, Moreno C, Noguera J. Hybrid notes cholecystectomy in an experimental model of laparoscopic acute cholecystitis. Surg Laparosc Endosc Percutan Tech. 2011 Apr;21(2):e65-9. doi: 10.1097/SLE.0b013e31820a2079. PMID 21471782
- [Background] Noguera JF, Cuadrado A, Sanchez-Margallo FM, Dolz C, Asencio JM, Olea JM, Morales R, Lozano L, Vicens JC. Emergency transvaginal hybrid natural orifice transluminal endoscopic surgery. Endoscopy. 2011 May;43(5):442-4. doi: 10.1055/s-0030-1256042. Epub 2010 Dec 16. PMID 21165824
- [Background] Noguera J, Dolz C, Cuadrado A, Olea J, Vilella A, Morales R. Hybrid transvaginal cholecystectomy, NOTES, and minilaparoscopy: analysis of a prospective clinical series. Surg Endosc. 2009 Apr;23(4):876-81. doi: 10.1007/s00464-008-0288-z. Epub 2009 Jan 1. PMID 19118420
- [Derived] Noguera J, Tejada S, Tortajada C, Sanchez A, Munoz J. Prospective, randomized clinical trial comparing the use of a single-port device with that of a flexible endoscope with no other device for transumbilical cholecystectomy: LLATZER-FSIS pilot study. Surg Endosc. 2013 Nov;27(11):4284-90. doi: 10.1007/s00464-013-3044-y. Epub 2013 Jun 29. PMID 23812286